CLINICAL TRIAL: NCT06054386
Title: Mobile-based Attentional Bias Modification Training (ABMT) for Socially Anxious Individuals
Brief Title: Attention Bias Modification Training for Social Phobia (ABMSP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWM 21.197
Record Dates: First submitted 2023-08-21; First posted 2023-09-26 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Social Anxiety Disorder
Keywords: Attentional bias; Cognitive process; Mobile training
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated ABM (I-ABM) (Active Comparator): The I-ABM will include four progressively difficult levels of training blocks, each containing 72 trials. Participants will be required to tap or swipe the probe in the correct direction during the first and second levels of training. The inhibitory control components will be included in the third and fourth levels, where participants should not respond to the probe under certain conditions. Each training will take 10-15 minutes, and participants will complete the sessions three times a week for three weeks.
  Interventions: Other: Attentional Bias Modification Training (ABMT)
- Placebo Training (PLT) (Placebo Comparator): The PLT has four training blocks that follow the same basic design as the I-ABM training. However, the PLT will not aim to change social anxiety-related attention bias. Participants will simply swipe or tap the probe regardless of the stimuli condition, which is expected to exert a minimum level of effect on changing the attention bias linked to social anxiety. Participants will complete the training three times per week for three weeks.
  Interventions: Other: General Attention Control Training

INTERVENTIONS:
Other: Attentional Bias Modification Training (ABMT) — The ABMT is aimed to modify attentional bias for negative stimuli in social anxiety by deliberately inducing the participant's attention to positive or neutral stimuli. In the training, after a pair of facial stimuli (e.g., threatening-neutral, neutral-neutral) are presented, a left or right arrow appears in one of the location. Participants are instructed to press the button in the correct direction as quickly and accurately as possible.
  Arms: Integrated ABM (I-ABM)
Other: General Attention Control Training — The general attention control training aimed to improve participants' general attention control ability by asking them to press a left or right arrow in the correct direction. The basic design of attention control training is the same as the ABMT, but the attention control training does not aim to alter the direction of attention toward or away from certain stimuli.
  Arms: Placebo Training (PLT)

SUMMARY:
Attentional bias has primarily been investigated as a primary cognitive etiology of social anxiety symptoms. Previous research has found that individuals with high social anxiety showed facilitated attentional engagement to threat stimuli or delayed disengagement of attention from threat. Attentional Bias Modification Training (ABMT) was developed through applying the attentional mechanism in social anxiety. During ABMT, participants are deliberately induced to shift their attention away from threat stimuli and toward neutral stimuli. Despite its proven effectiveness, a recent meta-study found that the effect size of ABMT is significant but too small. As a result, the current study focuses on improving the existing ABMT by incorporating integrative factors into attention training. The current study aims to integrate bottom-up and top-down cognitive processes in ABMT. Participants will be randomly assigned to one of two conditions (active or placebo training) and will complete the ABMT for three weeks. The ABMT's efficacy will be assessed by comparing pre- and post-training measures.

DETAILED DESCRIPTION:
Individuals with at least mild level of social anxiety symptoms will be invited to the current study. Participants will be randomly assigned to one of the two attention training conditions: a Integrated Attentional Bias Modification (I-ABM) training or placebo training (PLT). Before and after the training, participants will complete computerized tasks (e.g., attention network task, dot-probe task) and self-report questionnaires.

The basic design of I-ABM training will follow the dot-probe task, which will ask participants to swipe or tap on the probe in the correct direction. The I-ABM training aims to shift attention away from threatening stimuli or improve the inhibitory control ability. The PLT training will have the same basic design, but this will not include therapeutic components. Participants will complete the training three times per week for three weeks (a total of 9 training sessions), and there will be post-training and a 2-week follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of social anxiety disorder (based on the DIAMOND interview - Social anxiety module)
* Moderate or severe symptoms of social anxiety as revealed by the Liebowitz Social Anxiety Scale (LSAS score of ≥ 40) or MINI-SPIN (Score of ≥ 6)
* Ages 18-60
* English as a primary language
* Possession of a mobile device for access to the app (Inquisit 6)

Exclusion Criteria:

* Self-reported visual impairment that cannot be adjusted and will prevent them from clearly recognizing words and pictures on mobile screen
* Self-reported history of a bipolar disorder or psychotic disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mini-Social Phobia Inventory (Mini-SPIN) across Pre-training, Post-training, and 2-week follow up | Pre-training (before the first mobile training), Post-training (after three weeks of training), 2-Week follow-up (two weeks after the post training assessment)
  The Mini-Social Phobia Inventory (Mini-SPIN; Connor et al., 2001) is a 3-item measure which assesses the degree to which an individual experiences fear or avoidance in social situations. The measure uses a 5-point-Likert rating scale ranges from 0="not at all" to 4="extremely", with a total score range of 0-12. At a cutoff score of 6, the Mini-SPIN showed sensitivity of 89% and specificity of 90% for detecting generalized social anxiety disorder (Connor et al., 2001). The higher the scores, the more severe the symptoms of social anxiety.

SECONDARY OUTCOMES:
Change in Depression, Anxiety, and Stress Scale (DASS-21) across Pre-training, Post-training, and 2-week follow-up | Pre-training (before the first mobile training), Post-training (after three weeks of training), 2-Week follow-up (two weeks after the post training assessment)
  The Depression, Anxiety, and Stress scale (DASS-21; Lovibond & Lovibond, 1995) comprises 21 items with three subscales (depression, anxiety, and stress), each subscale consisting of seven items. Items are rated on a 4-point scale ranging from 0="did not apply to me at all" to 3="applied to me very much or most of the time". Total scores in each subscale are calculated by adding the scores from seven items and multiplying by two, with each subscale having a total score range of 0-42. The DASS-21 showed good internal reliability (coefficient alpha ranged between 0.74 and 0.93). The higher the scores, the more severe the depression, anxiety, and stress symptoms.
Change in Liebowitz Social Anxiety Scale (LSAS-SR) across Pre-training, Post-training, and 2-week follow-up | Pre-training (before the first mobile training), Post-training (after three weeks of training), 2-Week follow-up (two weeks after the post training assessment)
  The Liebowitz Social Anxiety Scale-Self Report (LSAS-SR; Liebowitz, 1987) assesses the severity of social anxiety and its associated avoidance across a variety of life domains. The LSAS-SR consists of 24 items that are rated on a 5-point scale from 0 ("none") to 4 ("very severe"). The LSAS-SR is divided into two subscales: fear and avoidance, with total scores ranging from 0-72 for each. The The higher the scores, the more severe the symptoms of social anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Han-Joo Lee, PhD, Principal Investigator — 414-229-5858
Locations (1):
- University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Amir N, Bomyea J, Beard C. The effect of single-session interpretation modification on attention bias in socially anxious individuals. J Anxiety Disord. 2010 Mar;24(2):178-82. doi: 10.1016/j.janxdis.2009.10.005. Epub 2009 Oct 27. PMID 19926442
- [Background] Connor KM, Kobak KA, Churchill LE, Katzelnick D, Davidson JR. Mini-SPIN: A brief screening assessment for generalized social anxiety disorder. Depress Anxiety. 2001;14(2):137-40. doi: 10.1002/da.1055. PMID 11668666
- [Background] Heeren A, Mogoase C, Philippot P, McNally RJ. Attention bias modification for social anxiety: A systematic review and meta-analysis. Clin Psychol Rev. 2015 Aug;40:76-90. doi: 10.1016/j.cpr.2015.06.001. Epub 2015 Jun 6. PMID 26080314
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Mogg K, Bradley BP. Selective orienting of attention to masked threat faces in social anxiety. Behav Res Ther. 2002 Dec;40(12):1403-14. doi: 10.1016/s0005-7967(02)00017-7. PMID 12457635
- [Background] Schofield CA, Johnson AL, Inhoff AW, Coles ME. Social anxiety and difficulty disengaging threat: evidence from eye-tracking. Cogn Emot. 2012;26(2):300-11. doi: 10.1080/02699931.2011.602050. Epub 2011 Oct 5. PMID 21970428
- [Background] Liebowitz MR. Social phobia. Mod Probl Pharmacopsychiatry. 1987;22:141-73. doi: 10.1159/000414022. No abstract available. PMID 2885745